CLINICAL TRIAL: NCT05430945
Title: Clinical Trial for the Safety and Efficacy of BCMA-targeted CAR-T Cells Therapy for Refractory/Relapsed Multiple Myeloma
Brief Title: A Study of BCMA-targeted CAR-T Cells Therapy for Refractory/Relapsed Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCMA-ZhejiangU
Record Dates: First submitted 2022-06-18; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: multiple myeloma; CAR T-cell therapy; BCMA
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of BCMA Targeted CAR T-cells (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: BCMA Targeted CAR T-cells

INTERVENTIONS:
Biological: BCMA Targeted CAR T-cells — Each subject receive BCMA Targeted CAR T-cells by intravenous infusion
  Other Names: BCMA Targeted CAR T-cells injection

SUMMARY:
Clinical Trial for the safety and efficacy of BCMA-targeted CAR-T cells therapy for refractory/relapsed multiple myeloma

DETAILED DESCRIPTION:
In this study, 100 patients with relapsed refractory multiple myeloma were proposed to undergo BCMA CAR-T cell therapy. Under the premise that its safety has been clarified in previous studies, further observation and evaluation of the effectiveness of BCMA CAR-T cell therapy for relapsed refractory multiple myeloma; At the same time, on the basis of expanding the sample size, more safety data on BCMA CAR-T cell treatment for relapsed refractory multiple myeloma were accumulated, including rare and delayed complications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed diagnosis of multiple myeloma (MM):

  1. Patients with BCMA positive relapsed/refractory MM;
  2. Relapsed after hematopoietic stem cell transplantation;
  3. Cases with recurrent positive minimal residual disease;
  4. Repeated MRD(+) refractory resistant cases
  5. Extramedullary leision which is hard to be eradicated by chemotherapy or radiotherapy.

     2. Anticipated survival time more than 12 weeks; 3. Transplant patients, regardless of their previous treatment, are eligible after relapse; 4. Those who voluntarily participated in this trial and provided informed consent.

     Exclusion Criteria:
* Subjects with any of the following exclusion criteria were not eligible for this trial:

  1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
  2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
  3. Pregnant (or lactating) women;
  4. With a graft-versus-host response, immunosuppressants are required;
  5. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
  6. Active infection of hepatitis B virus or hepatitis C virus;
  7. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
  8. Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
  9. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
  10. Other uncontrolled diseases that were not suitable for this trial;
  11. Patients with HIV infection;
  12. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after BCMA targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after BCMA targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Overall response rate (ORR) | At Day 28
  Assessment of ORR at Day 28
Overall survival (OS) | At Month 6, 12, 24
  Assessment of OS at Month 6, 12, 24
Quality of life(EORTC QLQ-C30) Core 30 (EORTC QLQ-C30) | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Hospital Anxiety and Depression Scale (HADS) score at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Medical College, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen R, Jin C, Liu K, Zhao M, Yang T, Zhang M, Xiao P, Feng J, Hong R, Fu S, Cui J, Huang S, Wei G, Huang H, Hu Y. Predictive value of pre-treatment circulating tumor DNA genomic landscape in patients with relapsed/refractory multiple myeloma undergoing anti-BCMA CAR-T therapy: Insights from tumor cells and T cells. Chin Med J (Engl). 2024 Nov 6;138(19):2481-90. doi: 10.1097/CM9.0000000000003306. Online ahead of print. PMID 39501801
- [Derived] Zhou L, Fu W, Wu S, Xu K, Qiu L, Xu Y, Yan X, Zhang Q, Zhang M, Wang L, Hong R, Chang AH, Yu J, Fu S, Kong D, Li L, Wang Y, Li Z, Jiang H, Huang J, Liu Z, Su N, Wei G, Hu Y, Huang H. Derivation and validation of a novel score for early prediction of severe CRS after CAR-T therapy in haematological malignancy patients: A multi-centre study. Br J Haematol. 2023 Aug;202(3):517-524. doi: 10.1111/bjh.18873. Epub 2023 May 16. PMID 37192741